CLINICAL TRIAL: NCT05225948
Title: Effects of Remote Ischemic Conditioning on Dynamic Cerebral Autoregulation, Blood Pressure and Heart Rate Variability in Patients With Cerebral Small Vessel Disease
Acronym: ESCAPE-SVD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESCAPE-SVD
Record Dates: First submitted 2021-12-09; First posted 2022-02-07 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Cerebral Small Vessel Diseases
MeSH Terms: conditions — Cerebral Small Vessel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC+Standard medical treatment (Active Comparator): Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflations of a blood pressure cuff to 200 mmHg. RIC will be conducted twice daily during the period of hospitalization. Besides, the patients will be treated with standard medical treatment according to consensus on diagnosis and treatment of cerebral small vessel disease in China 2015, including antiplatelet aggregation and lipid-stabilizing drugs as well as neurotrophic and circulation improving treatment.
  Interventions: Procedure: Remote ischemic conditioning
- Sham RIC+Standard medical treatment (Placebo Comparator): Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflations of a blood pressure cuff to 60 mmHg. RIC will be conducted twice daily during the period of hospitalization. Besides, the patients will be treated with standard medical treatment according to consensus on diagnosis and treatment of cerebral small vessel disease in China 2015, including antiplatelet aggregation and lipid-stabilizing drugs as well as neurotrophic and circulation improving treatment.
  Interventions: Procedure: Sham remote ischemic conditioning

INTERVENTIONS:
Procedure: Remote ischemic conditioning — Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflations of a blood pressure cuff to 200 mmHg. RIC will be conducted twice daily during the period of hospitalization.
  Arms: RIC+Standard medical treatment
Procedure: Sham remote ischemic conditioning — Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflations of a blood pressure cuff to 60 mmHg. RIC will be conducted twice daily during the period of hospitalization.
  Arms: Sham RIC+Standard medical treatment

SUMMARY:
The purpose of this study is to determine effects of remote ischemic conditioning on dynamic cerebral autoregulation, blood pressure and heart rate variability in patients with cerebral small vessel disease.

DETAILED DESCRIPTION:
In this study, 100 cases of cerebral small vessel disease in the First Hospital of Jilin University are divided into 2 groups according to the intention of the individual. On the basis of standard medical treatment, the experimental group receive in-hospital remote ischemic conditioning treatment for 200 mmHg, 2 times per day; the control group receive remote ischemic conditioning for 60 mmHg, 2 times per day during the period of hospitalization. Patients in both groups undergo several dynamic cerebral autoregulation and beat-to-beat monitoring respectively at baseline, 3-4 days of remote ischemic conditioning and the time the last in-hospital remote ischemic conditioning performed. Two groups will be followed up for 90 days to evaluate the effects of remote ischemic conditioning therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1) Regardless of age, sex;
* 2) Patients are diagnosed with cerebral small vessel disease, and neuroimaging shows new subcortical lacunar infarction (in line with one of the following):

  ① MRI examination Diffusion-weighted imaging (DWI) phase shows high signal intensity [Apparent Diffusion Coefficient (ADC) diffusion restriction] lesions < 20 mm diameter in subcortical, basal ganglia or brainstem , with or without corresponding clinical symptoms;

  ② With new clinical symptoms, MRI examination FLAIR sequence shows corresponding FLAIR high signal intensity lesions [diameter < 20 mm]) in subcortical, basal ganglia or pons;
* 3) Remote ischemic conditioning can be started within 7 days from onset;
* 4) Willing to participate and sign the informed consent.

Exclusion Criteria:

* 1) Vascular stenosis > 50% by Transcranial Doppler (TCD);
* 2) Previous history of intracranial hemorrhage or major bleeding in other parts of the body;
* 3) Previous history of atrial fibrillation or myocardial infarction within 6 months;
* 4) Moyamoya disease or hereditary cerebral small vessel disease, such as mitochondrial encephalopathy, CADASIL or Fabry;
* 5) The patients who had clear non-vascular white matter lesions, such as multiple sclerosis, adult white matter dysplasia, metabolic encephalopathy;
* 6) Severe hepatic and renal diseases, cancer or other major diseases related to medical and surgical procedures;
* 7) The patients who had the contraindication of remote ischemic conditioning treatment, such as severe soft tissue injury, fracture or vascular injury in the upper limb; Acute or subacute venous thrombosis, arterial occlusive disease, subclavian steal syndrome, etc;
* 8) Significant coagulation abnormalities;
* 9) Pregnant or lactating women;
* 10) The patients with disturbance of consciousness or agitation who cannot cooperate to dynamic cerebral autoregulation monitoring or beat-to-beat blood pressure monitoring;
* 11) Previous remote ischemic conditioning therapy or similar treatment;
* 12) Unwilling to be followed up or treated for poor compliance;
* 13) He/She is participating in other clinical research or has participated in other clinical research or has participated in this study within 3 months prior to admission;
* 14) Other conditions that the researchers think are not suitable for the group.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-30 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Phase Difference(PD) in Degree | within 7 days of RIC
  PD is a dynamic cerebral auto-regulation parameter derived from transfer function analysis.
Differences of blood pressure variability (BPV) in Degree after in-hospital remote ischemic conditioning finished between two groups | within 7 days of RIC
  BPV is defined as blood pressure oscillations in relation to the mean values.
Differences of heart rate variability (HRV) in Degree after in-hospital remote ischemic conditioning finished between two groups | within 7 days of RIC
  HRV is defined as heart rate oscillations in relation to the mean values.

SECONDARY OUTCOMES:
Differences of BPV in Degree after 3-4 days remote ischemic conditioning treatment between two groups | 3-4 days after RIC
  BPV is defined as blood pressure oscillations in relation to the mean values.
Differences of HRV in Degree after 3-4 days remote ischemic conditioning treatment between two groups | 3-4 days after RIC
  HRV is defined as heart rate oscillations in relation to the mean values.
PD in Degree | 3-4 days after RIC
  PD is a dynamic cerebral auto-regulation parameter derived from transfer function analysis.
Differences in modified Rankin Scale (mRS) Score between two groups | 3 months
  Modified Rankin Scale (mRS) Score ranged from 0 to 6, a low value represents a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China